CLINICAL TRIAL: NCT00889382
Title: A Phase 1/2 Study Evaluating Intermittent and Continuous OSI-906 and Weekly Paclitaxel in Patients With Recurrent Epithelial Ovarian Cancer (and Other Solid Tumors)
Brief Title: A Study Evaluating Intermittent and Continuous OSI-906 and Weekly Paclitaxel in Patients With Recurrent Epithelial Ovarian Cancer (and Other Solid Tumors)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSI-906-202; 2009-010319-34 (EudraCT Number)
Record Dates: First submitted 2009-04-06; First posted 2009-04-28 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer; Solid Tumors
Keywords: Ovarian; IGF-1R; Paclitaxel; Ovarian Cancer; OSI-906; Solid Tumors
MeSH Terms: conditions — Ovarian Neoplasms; Insulin-Like Growth Factor I, Resistance To | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase 1 Arm A (Experimental): Intermittent OSI-906 Once Daily (QD) on Days 1 - 3, 8 - 10, and 15 - 17 with paclitaxel on Days 1, 8, and 15 (except Treatment Period 1 (TP 1); in TP 1 OSI-906 on Days 1 - 3, 8 - 10, 15 - 17, and 22 - 24 with paclitaxel on Days 8, 15, and 22)
  Interventions: Drug: OSI-906; Drug: Paclitaxel
- Phase 1 Arm B1 (Experimental): Continuous OSI-906 Twice Daily (BID) (Days 1 - 21) with paclitaxel dosing on Days 1, 8, and 15;(except TP 1; in TP 1 OSI-906 on Days 1 - 3, 8 - 10, 15 - 17, and 22 - 24 with paclitaxel on Days 8, 15 and 22)
  Interventions: Drug: OSI-906; Drug: Paclitaxel
- Phase 1 Arm B2 (Experimental): Continuous OSI-906 BID (Days 1 - 21) with paclitaxel dosing on Days 1, 8, and 15 (except TP 1; in TP 1 OSI-906 on Days 1 - 3, 8 - 10, 5 - 17, and 22 - 24 with paclitaxel on Days 8, 15, and 22); (additional PK sampling on Days 9 or 13 0r 14 for TP 1)
  Interventions: Drug: OSI-906; Drug: Paclitaxel
- Phase 1 Arm B3 (Experimental): Continuous OSI-906 BID (Days 1 - 21) with paclitaxel dosing on Days 1, 8, and 15 with no separation in OSI-906 and paclitaxel dosing (except TP 1; in TP 1 continuous OSI-906 dosing 2 hours prior to the initiation of paclitaxel infusion on Day 8 only, with paclitaxel on Days 8, 15, and 22, and additional PK sampling on Day 9 or 13 or 14)
  Interventions: Drug: OSI-906; Drug: Paclitaxel
- Phase 2 Arm A (Experimental): Intermittent OSI-906 QD on Days 1 - 3, 8 - 10, and 15 - 17 with paclitaxel on Days 1, 8, and 15
  Interventions: Drug: OSI-906; Drug: Paclitaxel
- Phase 2 Arm B (Experimental): Continuous OSI-906 BID from Day 1 onwards with paclitaxel on Days 1, 8, and 15
  Interventions: Drug: OSI-906; Drug: Paclitaxel
- Phase 2 Arm C (Experimental): Paclitaxel on Days 1, 8, and 15
  Interventions: Drug: Paclitaxel
- Phase 2 Arm C Roll-over (Experimental): Continuous OSI-906 BID from Day 1 onwards
  Interventions: Drug: OSI-906

INTERVENTIONS:
Drug: OSI-906 — Administered orally
  Arms: Phase 1 Arm A; Phase 1 Arm B1; Phase 1 Arm B2; Phase 1 Arm B3; Phase 2 Arm A; Phase 2 Arm B; Phase 2 Arm C Roll-over
Drug: Paclitaxel — Administered intravenously
  Arms: Phase 1 Arm A; Phase 1 Arm B1; Phase 1 Arm B2; Phase 1 Arm B3; Phase 2 Arm A; Phase 2 Arm B; Phase 2 Arm C

SUMMARY:
This is a multi-center, randomized, open-label, phase 1/2 study of continuous weekly paclitaxel and escalating doses of intermittent or continuous OSI-906 in patients with recurrent/relapsed ovarian and other solid tumors.

DETAILED DESCRIPTION:
The phase 1 dose escalation portion will establish the maximum tolerated dose (MTD) in patients with advanced solid tumors. Once the recommended phase 2 dose (RP2D) is established for both schedules, the phase 2 study will begin. Patients with relapsed/recurrent epithelial ovarian cancer will be randomized 1:1:1 to 3 treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed epithelial ovarian carcinoma Patients with fallopian or peritoneal cancer will also be eligible
* Patients with any solid tumor that may be treated with weekly paclitaxel will be eligible for the phase 1 portion
* For the phase 2 portion, patients must have elevated CA125 levels evaluable/assessable according to Gynecological Cancer Intergroup (GCIG) criteria (ie, > 70 U/mL) documented by 2 measurements at least 1 week apart
* Patients must have radiologically confirmed progressive disease by RECIST v1.1 criteria within 6 months prior to randomization. (patients must have measurable disease according to RECIST v1.1)
* Eastern Cooperative Oncology Group (ECOG) performance status(PS) 0 -1
* Predicted life expectancy ≥ 12 weeks
* Patients may have had prior therapy, providing the following conditions are met:

  * Chemotherapy: Prior chemotherapy must have been completed at least 3 weeks prior to study enrollment (6 weeks for mitomycin C, nitrosoureas or high-dose carboplatin [≥ 600 mg/m²]and 4 weeks for investigational drugs

    1. Patient should have recovered from any drug-related toxicities (with the exception of grade 1 neuropathy and or alopecia)
    2. Phase 1: While there is no limit on the number of prior regimens for patients entered into the phase 1 portion, any prior taxane therapy must have been administered on a 3 week schedule
    3. Phase 2: Patients must have received prior chemotherapy, which must have contained a platinum and a taxanes at some point. Any prior taxanes therapy must have been administered on a 3 week schedule. A maximum of 2 prior chemotherapy regimens are permitted. Patients must be refractory radiologically confirmed by computerized tomography (CT) scan progressive disease (PD) during chemotherapy) or resistant (radiologically confirmed by CT scan PD within six months of completing chemotherapy) to their last platinum-containing chemotherapy regimen
  * Radiation: Patients may have had prior radiation therapy provided they have recovered from the acute, toxic effects of radiotherapy prior to registration/randomization. Radiated lesions cannot be chosen as the target lesions

    a. A minimum of 21 days must have elapsed between the end of radiotherapy and registration/randomization into the study unless the radiation affected less than 25% of bone marrow
  * Surgery: Previous surgery is permitted provided that adequate wound healing has occurred prior to registration/randomization
* Fasting glucose ≤ 150 mg/dL (8.3 mmol/L)
* Adequate hematopoietic, hepatic, and renal function defined as follows:

  * Neutrophil count ≥ 1.5 x 10 ^9 /L and platelet count > = 100 x 10^9/L;
  * Bilirubin ≤ 1.5 x Upper Limit of Normal (ULN);
  * AST and/or ALT ≤ 2.5 x ULN or < = 5 x ULN if patient has documented liver metastases; and
  * Serum creatinine ≤ 1.5 x ULN
* Female patient must be either:

  * Of non childbearing potential:

    1. post-menopausal (defined as at least 1 year without any menses) prior to Screening, or
    2. documented surgically sterile or status post hysterectomy (at least 1 month prior to Screening)
  * Or, if of childbearing potential:

    1. must have a negative urine pregnancy test at Screening, and
    2. must use two forms of birth control (one of which must be a barrier method) starting at Screening and throughout the study period and for 28 days [or 5 half lives, whichever is longer] after final study drug administration
* Female patient must not be breastfeeding at Screening or during the study period and for 28 days [or 5 half lives of the study drug whichever is longer] after final study drug administration
* Female patient must not donate ova starting at Screening and throughout the study period and for 28 days [or 5 half lives of the study drug whichever is longer] after final study drug administration
* Patients must provide verbal and written informed consent to participate in the study

Exclusion Criteria:

* Diabetes mellitus currently requiring medication (eg, insulin or oral hypoglycemics)
* During the phase 2 portion, patients with histology of abdominal adenocarcinoma of unknown origin or a diagnosis of a borderline ovarian tumor
* Previous or concurrent malignancies (excluding curatively treated basal or squamous cell carcinoma of the skin or cervical carcinoma in situ) unless the patient has been in remission for at least 3 years
* History of significant cardiovascular disease unless the disease is well-controlled. Significant cardiac diseases includes second/third degree heart block; significant ischemic heart disease; poorly controlled hypertension; congestive heart failure of New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea)
* History of cerebrovascular accident (CVA) within 6 months prior to registration/randomization or that is not stable
* Prior therapy with an insulin-like growth factor (IGF-1R) inhibitor
* Use of drugs that have a risk of causing QT interval prolongation within 14 days prior to Day 1 dosing
* Known or prior hypersensitivity to taxanes in spite of premedication or drugs containing Cremophor
* Gastro-intestinal abnormalities, including bowel obstruction, inability to take oral medication, requirement for intravenous (IV) alimentation,active peptic ulcer or prior surgical procedures or bowel resection affecting absorption
* Active infection or serious underlying medical condition (including any type of active seizure disorder within 12 months prior to registration/randomization) that would impair the ability of the patient to receive protocol treatment
* History of any psychiatric condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent
* Pregnancy or breast-feeding
* Symptomatic brain metastases that are not stable, require steroids, are potentially life threatening, or that have required radiation within 28 days prior to registration/randomization
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drug
* History of arrhythmia (multifocal premature ventricular contractions [PVCs], bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) that is symptomatic or requires treatment (≥ grade 3), left bundle branch block (LBBB), or asymptomatic sustained ventricular tachycardia are not allowed. Patients with atrial fibrillation controlled by medication are not excluded. Patients with mean QTcF interval ≥ 450 msec at screening are excluded
* Use of drugs that have a known risk of causing Torsade de Pointes (TdP) or that that have a risk of causing QT interval prolongation within 14 days prior to Day 1 dosing are prohibited
* Use of the potent CYP1A2 inhibitors ciprofloxacin and fluvoxamine. Other less potent CYP1A2 inhibitors/inducers are not excluded
* Participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half lives whichever is longer, prior to the initiation of Screening or during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2009-08-05 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2014-08-25 (Actual)

PRIMARY OUTCOMES:
Determine Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) | 28 days
  Primary outcome measure for Phase 1 portion
Progression Free Survival (PFS) | 36 months
  Primary outcome measure for the Phase 2 portion; The time from the date of randomization until date of radiographic disease progression per RECIST v1.1 or until death due to any cause

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 36 months
  The proportion of patients with a confirmed response of Complete Response (CR) or Partial Response (PR) per RECEIST v1.1
Cancer Antigen 125 (CA125) Response Rate | 36 months
  Response Rate is defined as at least 50% reduction in serum CA-125 levels from pretreatment levels; Response rate is the proportion of patients with a CA-125 response among evaluable patients
Duration of Response (DOR) | 36 months
  The time from the date of the first documented radiographic response (CR/PR) to first documented radiographic progression or death due to underlying cancer
Duration of CA-125 Response (CA-125 DOR) | 36 months
  The time from the date of the first documented CA-125 response to the date of CA-125 progression
Overall Survival (OS) | 36 months
  The time from the date of randomization until the documented date of death
Safety assessed via physician exam, vital signs, clinical laboratory tests, electrocardiograms (ECG), and adverse events | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator - Czech Republic, Principal Investigator — General Faculty Hospital, Charles University; Medical Director, Study Director — Astellas Pharma Global Development; Principal Investigator - Italy, Principal Investigator — Instituto Europeo de Oncologia
Locations (46):
- United States (8):
  - Mayo Clinic, Scottsdale, Arizona
  - Department of Obstetrics and Gynecology, University of California, Irvine, Orange, California
  - Horizon Oncology Center, Lafayette, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Blumenthal Cancer Center - Main, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
- Australia (9):
  - WestMead Hospital, Westmead, New South Wales
  - Mater Adult Hospital, South Brisbane, Queensland
  - Royal Adelaide Hospital, North Terrace, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Frankston Hospital, Frankston, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - St. John of God Hospital, Bunbury, Bunbury, Western Australia
  - Sir Charles Gairdner Hospital, Perth, Western Australia
  - St. John of Gog Hospital, Subiaco, Subiaco, Western Australia
- Canada (3):
  - Juravinski Cancer Center, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec
- Czechia (3):
  - University Hospital Hradec Kralove, Kralove
  - University Hospital Ostrava, Ostrava- Poruba
  - General University Hospital, Department of Obstetrics and Gynecology, Prague
- Italy (4):
  - Universitaria di Bologna Policlinico, Bologna
  - Ospedale di Carpi, AUSL di Modena, Carpi
  - Instituto Europeo di Oncologia, Milan
  - Oncology IDI- IRCSS, Roma
- Poland (3):
  - III Oddzial Onkologii Ginekologicznej, Lublin
  - Oddzial Radioterapii, Poznan
  - Klinika Onkologii AM w Poznaniu, Poznan
- Romania (4):
  - Institutul Oncologic Prof. Dr. Ion. Chiricuta Sectia de Oncologie Medicala, Cluj-Napoca
  - Institutul Oncologic Prof. Dr. Ion. Chiricuta Sectia Radiologie, Cluj-Napoca
  - Oncology Medical Centre SCM, Iași
  - Clinical Caunty Hospital Mures, Mures
- Russia (4):
  - Central Clinical Hospital, Moscow
  - Moscow City Oncology Hospital, Moscow
  - State Institution Medical Radiology Scientific Center, Obninsk
  - Sity Clinical Oncology, Saint Petersburg
- Ospedale San Giovanni, Bellinzona, Switzerland
- United Kingdom (7):
  - Drug Development Unit Royal Mardsen NHS Foundation Trust, Sutton, Surrey
  - Royal Marsden Hospital, London
  - University College Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Mount Vernon Cancer Center, Northwood
  - Churchill Hospital, Oxford
  - Christie NHS Foundation Trust, Withington

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=270